CLINICAL TRIAL: NCT05113901
Title: Methylprednisolone Taper to Treat Delayed Post-Operative Recovery After Total Knee Arthroplasty: a Double-Blind Randomized Controlled Trial
Brief Title: Medrol Dosepak Taper for Delayed Post-op Recovery After TKA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Extremely low participation, decided to focus on similar study instead
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Vasili Karas, Assistant Professor, Orthopedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 21080501
Record Dates: First submitted 2021-10-17; First posted 2021-11-09 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Total Knee Arthroplasty
Keywords: Methylprednisolone; Delayed recover; range of motion
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methylprednisolone taper (Active Comparator): 21 x 4mg tablets at 6 weeks, qualifying for MUA if ROM <90° at 8 weeks
  Interventions: Drug: Methylprednisolone
- Placebo taper (Placebo Comparator): 21 sugar tablets at 6 weeks with standard management, qualifying for MUA if ROM <90° at 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylprednisolone — 21 x 4mg tablets at 6 weeks, qualifying for MUA if ROM <90° at 8 weeks
  Arms: Methylprednisolone taper
Drug: Placebo — 21 sugar tablets at 6 weeks with standard management, qualifying for MUA if ROM <90° at 8 weeks
  Arms: Placebo taper

SUMMARY:
To evaluate the efficacy of a methylprednisolone taper on patients with decreased range of motion (ROM) or delayed recovery in the acute postoperative period following total knee arthroplasty (TKA).

Patients with decreased ROM or delayed recovery six weeks to three months post-TKA will improve ROM and patient-reported outcomes at two weeks post-treatment initiation of methylprednisolone taper, as compared to similar patients who receive a placebo taper.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most performed and efficacious orthopaedic procedures, with an estimated 7 million people living with a total knee prosthesis in 2010.1 The number of annual TKAs is predicted to increase by 85% by 2030 and 143% by 2050, equating to 1.26 million2 and 1.5 million3 procedures per year, respectively. In recent studies, knee prostheses have demonstrated their efficacy in 10-, 20-, and 25-year survival rates of 96.1%, 89.7%4, and 82.3%5, respectively. Similarly, comparing functional and patient-reported outcomes before and after surgery have confirmed the high success rate achieved with this procedure.6-10 However, recovery following total knee arthroplasty (TKA) in the acute postoperative period is variable. Most clinical improvements are achieved within the first three months postoperatively but can continue up to one year.11 There is currently a paucity of data evaluating the efficacy of oral corticosteroids in the six-week to three-month postoperative period in slowly recovering patients.

Few treatments have been studied for patients who fail to achieve early range of motion or pain reduction milestones in the perioperative period. Periarticular and systemic corticosteroids improve pain and function in the immediate postoperative period, without an increase in adverse events.12-16 Additional doses of corticosteroids administered at 24 and 48 hours postoperatively have demonstrated greater improvements in pain and ROM compared to perioperative administration, with no difference in complication rates.17-20 However, few studies have evaluated the use of oral corticosteroids within a multimodal pain management regimen. Gardiner et al. evaluated low-dose steroids 10 days immediately following lumbar laminectomy and/or discectomy, in addition to a standard opioid regimen, and reported decreased subjective pain scores.21 Gottshalk et al. reported decreased patient reported pain from postoperative days 4-7 in early published results of a randomized controlled trial investigating administration of a methylprednisolone taper immediately following distal radius repair.22 Importantly, the current literature demonstrates low- and short-dose corticosteroids are safe.23 Intraoperative corticosteroids have been shown to improve pain and function in the acute postoperative period, and additional doses in the immediate postoperative period can potentiate and prolong this beneficiary effect, without increasing adverse events. Therefore, a methylprednisolone taper six weeks post-TKA may benefit patients experiencing decreased ROM or delayed recovery, including residual pain.

Following TKA, care is taken to control pain, swelling, and stiffness, all of which may contribute to delayed recovery. For instance, more than 20% of TKA patients develop postoperative stiffness,24 known as arthrofibrosis, accounting for an estimated 28% of 90-day hospital readmissions.25 In treating patients with delayed recovery, corticosteroids are of particular interest because of its potent anti-inflammatory effect, evidenced by its ability to decrease postoperative levels of IL-6 and CRP.15 Corticosteroids block prostaglandin synthesis, which is responsible for sensitizing nociceptive pain receptors, and reduce vascular permeability, which causes edema following surgery.26, 27 Therefore, by reducing pain and edema, corticosteroids may allow for more effective physical therapy sessions and more rapid improvement in ROM and recovery following TKA.

To the best of our knowledge, this is the first study to investigate the utility of a methylprednisolone taper six weeks to three months postoperatively following TKA. The authors present a double-blinded, randomized-controlled trial evaluating the role of a methylprednisolone taper on patients with decreased ROM or delayed recovery in the acute postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary TKA with a diagnosis of osteoarthritis
* ≥ 18 years old
* ROM <90° by 3 weeks postoperatively without improvement to >90° by 6 weeks
* Requiring a 30-pill oxycodone refill
* NSAID allergy
* Thigh circumference discrepancy >2cm between legs from 3 to 6 weeks
* Defense and Veterans Pain Rating Scale (DVPRS) > 5 between 3 and 6 weeks
* Willingness to undergo randomization

Exclusion Criteria:

* Reported chronic corticosteroid or opiate use
* Suspected or confirmed periprosthetic joint infection
* Revision TKA
* Primary diagnosis other than osteoarthritis, including avascular necrosis, fracture, or post-traumatic arthritis
* American Society of Anesthesiologists (ASA) score ≥ 4
* Reported history of liver or renal disease
* Uncontrolled diabetes
* Immunosuppression
* ≤ 18 years old
* Inability to take oral medications
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Background] Maradit Kremers H, Larson DR, Crowson CS, Kremers WK, Washington RE, Steiner CA, Jiranek WA, Berry DJ. Prevalence of Total Hip and Knee Replacement in the United States. J Bone Joint Surg Am. 2015 Sep 2;97(17):1386-97. doi: 10.2106/JBJS.N.01141. PMID 26333733
- [Background] Sloan M, Premkumar A, Sheth NP. Projected Volume of Primary Total Joint Arthroplasty in the U.S., 2014 to 2030. J Bone Joint Surg Am. 2018 Sep 5;100(17):1455-1460. doi: 10.2106/JBJS.17.01617. PMID 30180053
- [Background] Bayliss LE, Culliford D, Monk AP, Glyn-Jones S, Prieto-Alhambra D, Judge A, Cooper C, Carr AJ, Arden NK, Beard DJ, Price AJ. The effect of patient age at intervention on risk of implant revision after total replacement of the hip or knee: a population-based cohort study. Lancet. 2017 Apr 8;389(10077):1424-1430. doi: 10.1016/S0140-6736(17)30059-4. Epub 2017 Feb 14. PMID 28209371
- [Background] Evans JT, Evans JP, Walker RW, Blom AW, Whitehouse MR, Sayers A. How long does a hip replacement last? A systematic review and meta-analysis of case series and national registry reports with more than 15 years of follow-up. Lancet. 2019 Feb 16;393(10172):647-654. doi: 10.1016/S0140-6736(18)31665-9. Epub 2019 Feb 14. PMID 30782340
- [Background] Callahan CM, Drake BG, Heck DA, Dittus RS. Patient outcomes following tricompartmental total knee replacement. A meta-analysis. JAMA. 1994 May 4;271(17):1349-57. PMID 8158821
- [Background] Ethgen O, Bruyere O, Richy F, Dardennes C, Reginster JY. Health-related quality of life in total hip and total knee arthroplasty. A qualitative and systematic review of the literature. J Bone Joint Surg Am. 2004 May;86(5):963-74. doi: 10.2106/00004623-200405000-00012. PMID 15118039
- [Background] Heath EL, Ackerman IN, Cashman K, Lorimer M, Graves SE, Harris IA. Patient-reported outcomes after hip and knee arthroplasty : results from a large national registry. Bone Jt Open. 2021 Jun;2(6):422-432. doi: 10.1302/2633-1462.26.BJO-2021-0053.R1. PMID 34182793
- [Background] Shan L, Shan B, Suzuki A, Nouh F, Saxena A. Intermediate and long-term quality of life after total knee replacement: a systematic review and meta-analysis. J Bone Joint Surg Am. 2015 Jan 21;97(2):156-68. doi: 10.2106/JBJS.M.00372. PMID 25609443
- [Background] Kane RL, Saleh KJ, Wilt TJ, Bershadsky B. The functional outcomes of total knee arthroplasty. J Bone Joint Surg Am. 2005 Aug;87(8):1719-24. doi: 10.2106/JBJS.D.02714. PMID 16085610
- [Background] Kagan R, Anderson MB, Christensen JC, Peters CL, Gililland JM, Pelt CE. The Recovery Curve for the Patient-Reported Outcomes Measurement Information System Patient-Reported Physical Function and Pain Interference Computerized Adaptive Tests After Primary Total Knee Arthroplasty. J Arthroplasty. 2018 Aug;33(8):2471-2474. doi: 10.1016/j.arth.2018.03.020. Epub 2018 Mar 17. PMID 29656980
- [Background] Deng Z, Li Y, Storm GR, Kotian RN, Sun X, Lei G, Gao S, Lu W. The efficiency and safety of steroid addition to multimodal cocktail periarticular injection in knee joint arthroplasty: a meta-analysis of randomized controlled trials. Sci Rep. 2019 May 7;9(1):7031. doi: 10.1038/s41598-019-43540-9. PMID 31065018
- [Background] Li Q, Mu G, Liu X, Chen M. Efficacy of additional corticosteroids to multimodal cocktail periarticular injection in total knee arthroplasty: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2021 Jan 22;16(1):77. doi: 10.1186/s13018-020-02144-0. PMID 33482865
- [Background] Mohammad HR, Hamilton TW, Strickland L, Trivella M, Murray D, Pandit H. Perioperative adjuvant corticosteroids for postoperative analgesia in knee arthroplasty. Acta Orthop. 2018 Feb;89(1):71-76. doi: 10.1080/17453674.2017.1391409. Epub 2017 Oct 25. PMID 29065753
- [Background] Yue C, Wei R, Liu Y. Perioperative systemic steroid for rapid recovery in total knee and hip arthroplasty: a systematic review and meta-analysis of randomized trials. J Orthop Surg Res. 2017 Jun 27;12(1):100. doi: 10.1186/s13018-017-0601-4. PMID 28655354
- [Background] Lex JR, Edwards TC, Packer TW, Jones GG, Ravi B. Perioperative Systemic Dexamethasone Reduces Length of Stay in Total Joint Arthroplasty: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Arthroplasty. 2021 Mar;36(3):1168-1186. doi: 10.1016/j.arth.2020.10.010. Epub 2020 Oct 16. PMID 33190999
- [Background] Backes JR, Bentley JC, Politi JR, Chambers BT. Dexamethasone reduces length of hospitalization and improves postoperative pain and nausea after total joint arthroplasty: a prospective, randomized controlled trial. J Arthroplasty. 2013 Sep;28(8 Suppl):11-7. doi: 10.1016/j.arth.2013.05.041. Epub 2013 Aug 9. PMID 23937923
- [Background] Kim JK, Ro DH, Lee HJ, Park JY, Han HS, Lee MC. Efficacy of Systemic Steroid Use Given One Day After Total Knee Arthroplasty for Pain and Nausea: A Randomized Controlled Study. J Arthroplasty. 2020 Jan;35(1):69-75. doi: 10.1016/j.arth.2019.08.026. Epub 2019 Aug 19. PMID 31563397
- [Background] Lei Y, Huang Z, Huang Q, Huang W, Pei F. Repeat Doses of Dexamethasone up to 48 Hours Further Reduce Pain and Inflammation After Total Hip Arthroplasty: A Randomized Controlled Trial. J Arthroplasty. 2020 Nov;35(11):3223-3229. doi: 10.1016/j.arth.2020.06.023. Epub 2020 Jun 17. PMID 32636109
- [Background] Xu H, Zhang S, Xie J, Lei Y, Cao G, Pei F. Multiple Doses of Perioperative Dexamethasone Further Improve Clinical Outcomes After Total Knee Arthroplasty: A Prospective, Randomized, Controlled Study. J Arthroplasty. 2018 Nov;33(11):3448-3454. doi: 10.1016/j.arth.2018.06.031. Epub 2018 Jul 4. PMID 30033064
- [Background] Gardiner D, McShane BJ, Kerr M, et al. Low-Dose Steroids to Decrease Postoperative Pain and Opioid Use. Journal for nurse practitioners. 2020;16(7):523-527. doi:10.1016/j.nurpra.2020.04.017
- [Background] Gottschalk M, Dawes A, Farley K, et al. Postoperative Methylprednisolone Taper Course for Distal Radius Fractures: Early Results of a Randomized Controlled Trial. Orthopaedic Proceedings; 2020:21
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Issa K, Banerjee S, Kester MA, Khanuja HS, Delanois RE, Mont MA. The effect of timing of manipulation under anesthesia to improve range of motion and functional outcomes following total knee arthroplasty. J Bone Joint Surg Am. 2014 Aug 20;96(16):1349-57. doi: 10.2106/JBJS.M.00899. PMID 25143495
- [Background] Schairer WW, Vail TP, Bozic KJ. What are the rates and causes of hospital readmission after total knee arthroplasty? Clin Orthop Relat Res. 2014 Jan;472(1):181-7. doi: 10.1007/s11999-013-3030-7. PMID 23645339
- [Background] Leppert W, Buss T. The role of corticosteroids in the treatment of pain in cancer patients. Curr Pain Headache Rep. 2012 Aug;16(4):307-13. doi: 10.1007/s11916-012-0273-z. PMID 22644902
- [Background] Vyvey M. Steroids as pain relief adjuvants. Can Fam Physician. 2010 Dec;56(12):1295-7, e415. PMID 21156893
- [Background] Prvu Bettger J, Green CL, Holmes DN, Chokshi A, Mather RC 3rd, Hoch BT, de Leon AJ, Aluisio F, Seyler TM, Del Gaizo DJ, Chiavetta J, Webb L, Miller V, Smith JM, Peterson ED. Effects of Virtual Exercise Rehabilitation In-Home Therapy Compared with Traditional Care After Total Knee Arthroplasty: VERITAS, a Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Jan 15;102(2):101-109. doi: 10.2106/JBJS.19.00695. PMID 31743238
- [Background] Guzik A, Druzbicki M, Wolan-Nieroda A, Turolla A, Kiper P. Estimating Minimal Clinically Important Differences for Knee Range of Motion after Stroke. J Clin Med. 2020 Oct 15;9(10):3305. doi: 10.3390/jcm9103305. PMID 33076214
- [Background] Research Programs. Accessed July 22, 2021. https://www.kneesociety.org/research-programs
- [Background] Huscher D, Thiele K, Gromnica-Ihle E, Hein G, Demary W, Dreher R, Zink A, Buttgereit F. Dose-related patterns of glucocorticoid-induced side effects. Ann Rheum Dis. 2009 Jul;68(7):1119-24. doi: 10.1136/ard.2008.092163. Epub 2008 Aug 6. PMID 18684744
- [Background] Saag KG, Koehnke R, Caldwell JR, Brasington R, Burmeister LF, Zimmerman B, Kohler JA, Furst DE. Low dose long-term corticosteroid therapy in rheumatoid arthritis: an analysis of serious adverse events. Am J Med. 1994 Feb;96(2):115-23. doi: 10.1016/0002-9343(94)90131-7. PMID 8109596
- [Background] Goldberg H, Firtch W, Tyburski M, Pressman A, Ackerson L, Hamilton L, Smith W, Carver R, Maratukulam A, Won LA, Carragee E, Avins AL. Oral steroids for acute radiculopathy due to a herniated lumbar disk: a randomized clinical trial. JAMA. 2015 May 19;313(19):1915-23. doi: 10.1001/jama.2015.4468. PMID 25988461
- [Background] Bartlett R, Hartle AJ. Routine use of dexamethasone for postoperative nausea and vomiting: the case against. Anaesthesia. 2013 Sep;68(9):892-6. doi: 10.1111/anae.12309. Epub 2013 Jul 15. No abstract available. PMID 23848377
- [Background] Feeley AA, Feeley TB, Feeley IH, Sheehan E. Postoperative Infection Risk in Total Joint Arthroplasty After Perioperative IV Corticosteroid Administration: A Systematic Review and Meta-Analysis of Comparative Studies. J Arthroplasty. 2021 Aug;36(8):3042-3053. doi: 10.1016/j.arth.2021.03.057. Epub 2021 Apr 24. PMID 33902983
- [Background] Sauerland S, Nagelschmidt M, Mallmann P, Neugebauer EA. Risks and benefits of preoperative high dose methylprednisolone in surgical patients: a systematic review. Drug Saf. 2000 Nov;23(5):449-61. doi: 10.2165/00002018-200023050-00007. PMID 11085349
- [Background] Dilisio MF. Osteonecrosis following short-term, low-dose oral corticosteroids: a population-based study of 24 million patients. Orthopedics. 2014 Jul;37(7):e631-6. doi: 10.3928/01477447-20140626-54. PMID 24992058
- [Background] Madanagopal SG, Kovaleski JE, Pearsall AW 4th. Survey of short-term oral corticosteroid administration by orthopaedic physicians in college and high school athletes. J Sports Sci Med. 2009 Mar 1;8(1):37-44. eCollection 2009. PMID 24150554

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methylprednisolone Taper | Placebo Taper
Started | 4 | 0
Completed | 3 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early, only 4 subjects were consented, none were randomized to the placebo by the time the study ended.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone Taper | Placebo Taper | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 63.31 [61.30 to 67.02] |  | 63.31 [61.30 to 67.02]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 0 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion in Degrees at Pre and Post Treatment
Description: Range of motion (ROM) from pre-treatment to six weeks following treatment. Patients started treatment after total knee replacement surgery and presented to clinic with at least one inclusion criteria to be enrolled. Range of motion in degrees is taken at each visit by a clinician (standard of care), starting at zero degrees (straight leg) to about 135 degrees. The ROM was documented as part of consenting and enrollment into study. Subjects returned to the office at 6 weeks post treatment where ROM was performed in a clinic setting once again and documented. ROM is done using a goniometer by a clinician in each clinic.
  This study was terminated early, therefore of the 4 enrolled, zero were randomized to the placebo group. Only 1 of the four subjects completed the 6 weeks, however, ROM was captured on all as standard of care.
Time Frame: Baseline, Week 6 Following Treatment
Population: **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: Range of Motion in Degrees
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
Range of Motion in Degrees
  Pre treatment | 82.5 [50 to 95] |
  Post treatment | 112 [105 to 120] |

2. Secondary Outcome: Patient Reported Outcome Measures: Post Treatment Pain Scores (6 Weeks)
Description: Using daily defense and veterans pain rating scale (DVPRS) on a scale of 1 to 10, 10 being the worst.
  Please note, only one patient made it to the 6 week post treatment mark of the 4 enrolled. The study was terminated and none of the patients were randomized to the placebo group. All other patients followed up but were not interested in continuing. No range could be provided given only one subject answered and completed this visit
Time Frame: 6 weeks post treatment
Population: This study was terminated early, only 1 of the 4 enrolled subjects reached the 6 week mark.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 1 | 0
score on a scale | 1.93 |

3. Secondary Outcome: Patient Reported Outcome Measures: Pre Treatment Pain Scores Using Knee Society Scores
Description: Knee society score (KSS); done standard of care on a scale of 0-100, where 100 means a more functional knee
  **Please note, the study was terminated early, only 4 subjects were enrolled and none were randomized to the placebo group.
Time Frame: pre treatment
Population: **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 66.25 [55 to 90] |

4. Secondary Outcome: Patient Reported Outcome Measures: Post Treatment Pain Scores
Description: Knee society score (KSS); done standard of care on a scale of 0-100, where 100 means a more functional knee.
  **Please note, the study was terminated early, only 4 subjects were enrolled and none were randomized to the placebo group. At 3 weeks post treatment, only 3 of the 4 subjects enrolled were still part of the study.
Time Frame: 3 weeks post treatment
Population: **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 3 | 0
score on a scale | 68.33 [60 to 85] |

5. Secondary Outcome: Patient Reported Outcome Measures: Post Treatment Pain Scores
Description: Knee society score (KSS); done standard of care on a scale of 0-100, where 100 means a more functional knee.
  **Please note, the study was terminated early, only 4 subjects were enrolled and none were randomized to the placebo group. This is a standard of care survey available on all subjects.
Time Frame: 6 weeks post treatment
Population: **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 3 | 0
score on a scale | 78.75 [55 to 90] |

6. Secondary Outcome: Patient Reported Outcome Measures:(Immediate) Post Treatment Pain Scores
Description: Using Daily Visual Analogue Scale (VAS) pain score, which measures intensity of pain on a scale of 0 (no pain) to 10 (worst pain possible).
  **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Time Frame: Days 1 through 6 following treatment
Population: **Please note, this study was terminated early, only enrolling 4 patients, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale
  Day 1 | 2.33 [0 to 4] |
  Day 2 | 3 [0 to 8] |
  Day 3 | 1.33 [0 to 3] |
  Day 4 | 1.33 [0 to 3] |
  Day 5 | 1.67 [1 to 3] |
  Day 6 | 2.3 [1 to 3] |

7. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee After Surgery and Treatment
Description: Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR), a survey given to patients standard of care containing 7 questions. The score ranges from 0 to 100 where zero represents total disability and 100 represents a perfect knee health.
Time Frame: pre treatment
Population: Please note, the study was terminated early and only 4 patients were enrolled. Of the 4 enrolled, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 50.04 [28 to 68.28] |

8. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee After Surgery and Treatment
Description: as for outcome 7
Time Frame: 6 weeks after treatment
Population: Please note, this study was terminated early where we only enrolled 4 subjects. Of the 4, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 72.12 [61.58 to 91.98] |

9. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee Before Treatment
Description: Veterans Rand 12-Item Health Survey (VR-12), a survey of 12 questions to measure health relating to patient's quality of life. Scored as summary of mental and physical, measure in standard deviations. The scale range is 0 to 100, where a score of 100 represents the best physical and mental health and zero is the worst outcome.
Time Frame: pre treatment
Population: as for outcome 8
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 38.73 [30.19 to 44.62] |

10. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee 6 Weeks After Treatment
Description: VR-12: Assesses physical functioning, physical/ mental limitations. Scored as summary of mental and physical, measure in standard deviations. The scale range is 0 to 100, where a score of 100 represents the best physical and mental health and zero is the worst outcome.
Time Frame: 6 weeks after treatment
Population: This study was terminated early after only 4 subjects were enrolled. None of these patients were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 50.28 [41.84 to 57.79] |

11. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee Before Treatment
Description: Single Assessment Numeric Evaluation (SANE), a single-question patient rating of 0-100, scoring their function to the area being treated. Zero represents a poor functional knee and 100 is the best functioning.
Time Frame: pre treatment
Population: Please note, this study was terminated early with only 4 patients enrolled. Of the 4 enrolled, none were randomized to the placebo group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 29.5 [0 to 55] |

12. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee 6 Weeks After Treatment
Description: as for outcome 11
Time Frame: 6 weeks after treatment
Population: as for outcome 11
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 89.5 [80 to 100] |

13. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee Prior to Treatment
Description: Forgotten Joint Score (FJS) is a survey scored ranging from 0 to 100, where a high score indicates a high degree of a forgetting they have an artificial joint, which is an ideal outcome.
Time Frame: pre treatment
Population: as for outcome 11
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 91.67 [75 to 100] |

14. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee 6 Wks After Treatment
Description: as for outcome 13
Time Frame: 6 weeks after treatment
Population: as for outcome 11
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 57.82 [47.92 to 66.67] |

15. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee Prior to Treatment
Description: UCLA activity score, on a scale of 1 to 10 where 10 is the most active patient with examples of activities
Time Frame: pre treatment
Population: as for outcome 11
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 4.25 [4 to 5] |

16. Secondary Outcome: Patient Reported Outcome Measures: Overall Assessment of Knee 6 Weeks After Treatment
Description: UCLA activity score, on a scale of 1 to 10 where 10 is the most active patient with examples of activities
Time Frame: 6 weeks after treatment
Population: as for outcome 11
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
score on a scale | 5.25 [4 to 6] |

17. Secondary Outcome: Number of Participants With Complications Following Treatment
Description: Manipulations under anesthesia (MUAs) following total knee arthroplasty surgery and treatment
Time Frame: within 90 days after initial total knee arthroplasty
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
Participants | 0 | 0

18. Secondary Outcome: Adverse Events or Outcomes Outside of Manipulations Under Anesthesia
Description: Adverse outcomes including infection, avascular necrosis, and 90-day readmission rates
Time Frame: within 90 days after initial total knee arthroplasty
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Methylprednisolone Taper | Placebo Taper
Number analyzed (Participants) | 4 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days following treatment
Description: Please note, this study was terminated early with only 4 patients enrolled. Of the 4 enrolled, none were randomized to the placebo group.
Arm/Group | Methylprednisolone Taper | Placebo Taper
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT05113901/Prot_SAP_001.pdf